CLINICAL TRIAL: NCT06051318
Title: Individual Effect of Diet on Postprandial Glycemic Response and Its Relationship with Gut Microbiome Profile in Healthy Subjects: Protocol for a Series of Randomized N-of-1 Trials
Brief Title: Relationship Between Individual Effect of Diet on Postprandial Glycemia and Gut Microbiome Profile in Healthy Subjects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BiomeHub Biotechnology Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 68325123.0.0000.5355
Record Dates: First submitted 2023-09-12; First posted 2023-09-22 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Glucose Metabolism Disorders; Health Behavior; Diabetes; Metabolic Disease
Keywords: Glycemic response; Precision nutrition; Gut Microbiome; Biomarkers; Sequencing analysis; N-of-1 trials
MeSH Terms: conditions — Glucose Metabolism Disorders; Health Behavior; Diabetes Mellitus; Metabolic Diseases

STUDY DESIGN:
Intervention Model Description: The study is a N-of-1 randomized series trial with multiple crossovers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standardized breakfast A (Experimental): Consumption order: Participants will initiate the interventional period by eating the low-carb muffin first following the established muffin order for the next days.
  Interventions: Other: Standardized breakfast A
- Standardized breakfast B (Experimental): Consumption order: Participants will initiate the interventional period by eating the vegan muffin first following the established muffin order for the next days.
  Interventions: Other: Standardized breakfast B

INTERVENTIONS:
Other: Standardized breakfast A — Participants will initiate the interventional period by eating the low-carb muffin first following the established muffin order for the next days.
  Arms: Standardized breakfast A
Other: Standardized breakfast B — Participants will initiate the interventional period by eating the vegan muffin first following the established muffin order for the next days.
  Arms: Standardized breakfast B

SUMMARY:
When all the food we eat is digested, it will increase blood glucose. Two people can have different glucose blood levels to the same food and one reason can be bacteria live in our gut. There are more than a thousand bacteria species in our gastrointestinal tract that have an important role in the proper functioning of our body, so our gut microbiome is a key piece for our nutrition and blood glucose control.

Nowadays, one of the major public health concerns is the rise of people with diabetes (a disease characterized by an increase in blood glucose) and the increase in obesity, in which one of several risks is diabetes. There are multiple reasons for people develop those diseases, however, some care on diet management can prevent, delay, or improve the effects of these illnesses. Therefore, this study proposes studying the blood glucose variation between healthy volunteers and if there is a relationship between that variation and the intestinal bacteria present. These results can help doctors and nutritionists elaborate a personalized diet for people who need blood glucose level control.

The investigators are recruiting volunteers aged 18 to 60, healthy, living at Florianopolis and the surroundings to participate in this crossover randomized N-of-1 study. The participants must collect fecal samples. After collection, the participants will meet the investigators and receive a kit containing ten standardized breakfasts, with two kinds of muffins, and a kit containing a glucose monitor (Abbott Freestyle Libre-CE marked) to monitor their blood sugar levels. The volunteers must have breakfast with the standardized meals and monitor the fasting glucose blood and postprandial glucose blood levels for ten consecutive days. Besides, they must take notes (like a diet diary) about all the food they ingest during the day in ten days of the study.

DETAILED DESCRIPTION:
Choice of design: The study is a N-of-1 randomized series trial with multiple crossovers.

Study population: This study will monitor healthy volunteers and they will be recruited via social media like Facebook, Instagram, and LinkedIn platforms.

Screening Assessment: The participants will be selected based on inclusion and exclusion criteria by study management researchers. Recruitment will be done via e-mail the participant will receive all the information about the study including the consent term and the anthropometric questionnaire. If he/she accepts it will be sent a collection kit for the fecal samples to the participant's address.

Study duration: Each participant will take part in the study for ten days. Dietary intervention: The participants will receive 10 standardized meals, divided into two kinds of muffins, which consist of a low-carbohydrate diet and a vegan one. The low-carb muffin will have a glycemic control characteristic, with a low carbohydrate content, below 45% of the carbohydrates recommended by the Acceptable Macronutrient Distribution Ranges (AMDR), while the vegan muffin will consist entirely of plant-based foods in the recommended macronutrient proportions. Both muffins will be similar in calories and standardized at 25% of daily calories, equivalent to the caloric distribution of breakfast.

After the fecal collection, the participant must introduce the standardized meals and the glucose monitoring device inserted. The meal order must obey the randomization established. Before breakfast, the participant will have to measure the fasting glucose with the monitoring glucose device and then eat the breakfast. After ingesting the muffin, the participant will measure glucose levels every 30 minutes over a 2-hour period, totaling four postprandial glucose measurements. Participants are free to eat whatever they wish at all other times, but they will report every meal in a diet diary. Together with breakfast, they can drink coffee without milk and sugar or water. The volunteers shouldn't do fasting exercises either for about two hours after breakfast.

Anthropometry dietary and lifestyle questionnaire: Before the participants initiate the intervention they will answer a simple questionnaire about their weight, height, gastrointestinal symptoms, stool shape, drugs in use, antibiotics, proton pump inhibitors use, any diagnosis of chronic disease, kind of diet, and activity information.

Digital devices: Participants will be asked to record daily dietary intake on an online platform, like Google Sheets. The continuous glucose monitor (Freestyle Libre, CGM) will be inserted on the back of the upper arm by themselves, or if they prefer it can be inserted by one of the researchers when they receive all the study kits. Subcutaneous interstitial fluid glucose will be measured before breakfast and two hours later. At the end of the intervention period, the CGM can be removed at home. Researchers' email addresses and cellphone number will be always available to participants to make any question.

Digital app: Participants will need to download the app FreeStyle LibreLink for the subcutaneous interstitial fluid glucose to be measured with their cellphones.

Sample size: The sample size was calculated through simulation, assuming a Gaussian multilevel model, comparing two diets with random intercept and diet effects per participant. The simulation assumptions were validated with a nutritionist to ensure plausible values for the outcome, intra-individual and inter-individual outcome variability, and individual effect variability. A minimum clinically significant effect on postprandial blood glucose of 15 mg/dL was determined. This value was used to define the expected range for 95% of true individual effects. The number of cycles was fixed at five to minimize the study time for each recruited participant. Under these assumptions, the simulation of 10,000 series of N-of-1 clinical trials determined it would be recruiting 80 participants.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 18.5 and < 30
* Willing to use an intradermal continuous glucose monitoring sensor during the 10-day study
* Own a mobile phone with NFC technology
* Willing to provide a fecal swab sample and a stool sample
* Understanding, agreement, and signing of the approved Informed Consent Form (ICF) by the Ethics Committee (CEP)

Exclusion Criteria:

* Pregnant or lactating women
* Diagnosis of any gastrointestinal disorder or disease (Irritable Bowel Syndrome, Ulcerative Colitis, Crohn's Disease)
* Intolerance or allergy to any diet ingredient
* Autoimmune disorder (Lupus, Type 1 Diabetes, Celiac Disease) or infectious disease
* Diabetes diagnosis
* Cancer diagnosis, acute myocardial infarction, or stroke in the last 6 months
* Use of hypoglycemic medication
* Use of proton pump inhibitors, immunosuppressants, or antimicrobials in the last 3 months
* Use of laxative medications in the last 30 days
* Underwent invasive procedures or surgery in the last 6 months
* Admission to ICU in the last 2 years
* Participation in any experimental study or ingestion of any experimental drug within twelve months prior to the start of this study, in accordance with RDC 251/97
* Inability to read and understand the informed consent form

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-06-06 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Fasting subcutaneous interstitial fluid glucose measured by continuous glucose monitor (CGM) | 0 min
  All participants will measure fasting subcutaneous interstitial fluid glucose before breakfast with CGM device during 10 days of intervention. The device measures subcutaneous interstitial glucose in the mg/dL unit and the reading is done through the device's app by cell phone approximation. Data is retained in the app and will be shared with researchers.
Postprandial subcutaneous interstitial fluid glucose measured by continuous glucose monitor (CGM) | 0 min
  All participants will measure postprandial subcutaneous interstitial fluid glucose every 30 minutes over two hours after breakfast with CGM device during 10 days of intervention. The device measures subcutaneous interstitial glucose in the mg/dL unit and the reading is done through the device's app by cell phone approximation. Data is retained in the app and will be shared with researchers.

SECONDARY OUTCOMES:
Participant's gut microbiome species richness | 2 weeks
  Gut microbiome profile will be performed by 16S sequencing from participant's fecal sample.

CONTACTS AND LOCATIONS:
Overall Officials: Caetana P. Zamparette, PhD, Study Chair — Researcher fellow; Bianca L. Teixeira, PhD, Study Chair — Clinical research; Giuliano Netto, Msc, Study Chair — Bioinformatics development and maintenance; Aline FR Sereia, PhD, Study Chair — Chief Operating Officer; Ana P. Christoff, PhD, Study Chair — Researcher R&D; Daniela C Bastiani, B.Sc, Study Chair — Laboratory manager; Fernanda RG Piazza, Msc, Study Chair — Nutricionist; Michele P Rode, PhD, Study Chair — Product Owner; Milene H Moraes, PhD, Study Chair — Researcher R&D; Natália M Gutierrez, Study Chair — Laboratory analyst; Luiz Felipe V. de Oliveira, PhD, Principal Investigator — BiomeHub CEO
Locations (1):
- BiomeHub, Florianópolis, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: No
We don't have a plan yet.